CLINICAL TRIAL: NCT02647112
Title: Utility of Bladder EpiCheck for Detection of Recurrent Urothelial Carcinoma A Multicenter, Prospective Blinded Study
Brief Title: Utility of Bladder EpiCheck for Detection of Recurrent Urothelial Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nucleix Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: UC-EpiCheck-EU-01
Record Dates: First submitted 2015-12-16; First posted 2016-01-06 (Estimated); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Bladder Cancer
Keywords: Bladder cancer; Urine; Methylation
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bladder EpiCheck (Experimental): Urine sample will be tested with the Bladder EpiCheck in conjunction with cystoscopy and cytology
  Interventions: Other: Bladder EpiCheck
- Practice of medicine (No Intervention): Practice of medicine including cystoscopy and cytology

INTERVENTIONS:
Other: Bladder EpiCheck — Urine test for the monitoring of bladder cancer recurrence
  Arms: Bladder EpiCheck

SUMMARY:
Clinical trial to determine the performance characteristics (sensitivity and specificity) of the Bladder EpiCheck test compared to the gold standard cystoscopy and pathology.

DETAILED DESCRIPTION:
Clinical trial to determine the performance characteristics (sensitivity and specificity) of the Bladder EpiCheck test compared to the gold standard cystoscopy and pathology in patients under monitoring for reccurrence of bladder cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with incident or recurrent urothelial cell carcinoma and undergoing surveillance monitoring for urothelial cell carcinoma
* Has all urothelial cell carcinoma tumor resected within the past 12 months
* Has a plan for cystoscopic surveillance

Exclusion Criteria:

* Planning to undergo radical cystectomy or chemotherapy-radiation for UCC

Ages: 22 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1050 (Actual)
Dates: Start 2015-12; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Sensitivity (the proportion of positives that are correctly identified as such by the gold standard) | Day 1
  the proportion of positives that are correctly identified as such by the gold standard
Specificity (the proportion of negatives that are correctly identified as such by the gold standard) | Day 1
  the proportion of negatives that are correctly identified as such by the gold standard

CONTACTS AND LOCATIONS:
Overall Officials: Shmulik Adler, Study Director — Nucleix Ltd.; Fred Witjes, Prof., Principal Investigator — Radboud University Medical Center
Locations (6):
- Tubingen University Medical Center, Tübingen, Germany
- Meir Medical Center, Kfar Saba, Israel
- Netherlands (3):
  - AMC Medical Center, Amsterdam
  - ZGT Medical Center, Hengelo
  - Radboud University Medical Center, Nijmegen
- Vall D'Hebron Medical Center, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No